CLINICAL TRIAL: NCT05314699
Title: The Order Effect of Acute Concurrent Exercise on Executive Function: An Event-Related Potential Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_rueihongli_CE_Order
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Executive Function
Keywords: acute exercise; concurrent exercise; inhibition; cognitive flexibility
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to three group, namely the resistance-aerobic exercise group (RA), the aerobic-resistance exercise group (AR), and the reading control group (RC). Participants in RA groups were asked to finish 5 min warm-up, 13 min resistance exercise, 12 min aerobic exercise, and 5 min cool down. Participants in AR groups were asked to finish 5 min warm-up, 12 min aerobic exercise, 13 min resistance exercise, and 5 min cool down. Participants in RC group were required to finish 35 min reading. All groups took a 30 min cognitive test before and after the intervention.The blood lactate were collected before, 17 minutes after, and after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- resistance-aerobic exercise group, RA (Experimental): Participants conduct 5-min warm up, 13-min resistance exercise, 12-min aerobic exercise, and 5-min cool down.
  Interventions: Behavioral: resistance-aerobic exercise, RA
- aerobic-resistance exercise group, AR (Experimental): Participants conduct 5-min warm up, 12-min aerobic exercise, 13-min resistance exercise, and 5-min cool down.
  Interventions: Behavioral: aerobic-resistance exercise, AR
- reading control group, RC (No Intervention): Participants conduct reading for 35 minutes.

INTERVENTIONS:
Behavioral: resistance-aerobic exercise, RA — Participants conduct 5-min warm up, 13-min resistance exercise, 12-min aerobic exercise, and 5-min cool down.
  Arms: resistance-aerobic exercise group, RA
Behavioral: aerobic-resistance exercise, AR — Participants conduct warm up for 5-min, aerobic exercise for 12-min, resistance exercise for 13-min, and 5-min cold down.
  Arms: aerobic-resistance exercise group, AR

SUMMARY:
Executive function is a high-level cognition which plays an important role in our life. Meta-analysis study has demonstrated that acute exercise could improve executive function. However, it is still unclear whether executive function can be enhanced by the concurrent exercise that combines aerobic and resistance exercise. Moreover, the sequence of concurrent exercise may result in different blood lactate concentration which may affect executive function. Therefore, the purposes of present study are: (1) Measuring the order effect of acute concurrent exercise on executive function. (2) Measuring whether order effect of acute concurrent exercise on executive function is mediated by blood lactate.

DETAILED DESCRIPTION:
Executive function is a high-level cognition which plays an important role in academic performance, career, and interpersonal relationship. Meta-analysis study has demonstrated that acute exercise could improve executive function, and also observed similar positive effect through both aerobic and resistance exercise. However, it is still unclear whether executive function can be enhanced by the concurrent exercise that combines aerobic and resistance exercise. Moreover, the sequence of concurrent exercise may result in different blood lactate concentration which may affect executive function. Therefore, the purposes of present study are: (1) Measuring the order effect of acute concurrent exercise on executive function. (2) Measuring whether order effect of acute concurrent exercise on executive function is mediated by blood lactate.

ELIGIBILITY:
Inclusion Criteria:

1. no history of psychiatric or neurological disorders
2. no history of cardiovascular disease
3. normal or corrected to normal vision and normal color perception
4. right handed
5. 18.5 < BMI < 27

Exclusion Criteria:

1. Diagnosed with epilepsy

Ages: 21 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Stroop test | 30 minutes
  The Stroop task consists of neutral, congruent, and incongruent trials. In neutral trials, colored rectangles were presented and participants were instructed to respond to whether the squares were red, blue, or green. For congruent and incongruent trials, participants were presented with the names of the three Chinese color words of 紅 (red), 藍 (blue), or 綠 (green) printed in either the same (congruent) or different (incongruent) ink color and instructed to respond to the color of the ink while inhibiting the meaning of the word.
task switch test | 30 minutes
  The shifting aspect of executive function was assessed by means of a computer version of the task-switching test. In brief, each participant was presented with six blocks of 64 trials. For the first block, the participant was required to identify whether the stimulus (i.e., digits 1-9, without digit 5) within the solid-line square was greater/less than the digit 5. For the second block, the participant identified whether the stimulus within the dotted-line square was even/odd. The blocks 3-6 consisted of an equal number of stimuli from the first and second blocks forming an alternating-runs paradigm.

OTHER OUTCOMES:
blood lactate | 1 minutes
  The lactic acid system is one of the important systems of human energy metabolism. In addition to supplying energy to muscles, it can also be used as an energy source for brain energy metabolism. When people doing exercise, the concentration of blood lactate will be increased, and the lactate acid system will replace the glucose system as the main energy source for the brain. In the present study, blood lactate were collected from fingertip with a lancet and measured by lactate analyzer before, 17 minutes after, and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No